CLINICAL TRIAL: NCT06961162
Title: A Prospective, Single-Center Study: Evaluation of Chronic Kidney Disease Severity Using Ultrasonic Viscoelastic Parameters Combined With Clinical Indicators-With Histopathological Results as Gold Standard
Brief Title: The Accuracy of Ultrasonic Viscoelastic Imaging in Evaluating the Severity of Chronic Kidney Diseases
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2023736
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease(CKD)
Keywords: chronic kidney disease; sonoelastogrphy; fibrosis; inflammation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Fibrosis; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the role of ultrasonic viscoelastic parameters in the assessing the severity of chronic kidney disease. The main question it aims to answer is:

The accuracy of ultrasonic viscoelastic parameters in evaluating the degree of renal fibrosis and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* (1) fulfilled the diagnostic criteria for CKD (disease course > 3months); (2) underwent renal biopsy, (3) a prior 2D-SWE evaluation preceding the renal biopsy, and (4) obtained informed written consent.

Exclusion Criteria:

* (1) the presence of multiple renal cysts, calculi, hydronephrosis, or masses that could potentially interfere with the analysis conducted through 2D-SWE: (2) unsuccessful 2D-SWE measurements ;(3) biopsy specimens deemed inadequate due to insufficient length (less than 10 mm) or fewer than 10 glomeruli, and (4) incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CKD patients who underwent renal biopsy at Peking University Third Hospital based on clinical requirements
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
renal fibrosis degree | one week

CONTACTS AND LOCATIONS:
Overall Officials: Ligang Cui, Dr, Principal Investigator — Department of Ultrasound, Peking University Third Hospital
Locations (1):
- Department of Ultrasound, Peking University Third Hospital, Beijing, Beiing, China

IPD SHARING:
Plan to Share IPD: No